CLINICAL TRIAL: NCT05624840
Title: Safety and Clinical and Virologic Outcomes in COVID-19 Patients With Chronic Kidney Disease Treated With Nirmatrelvir-ritonavir
Brief Title: Safety and Clinical and Virologic Outcomes in CKD Patients Treated With Nirmatrelvir-ritonavir
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Consultant, Chinese University of Hong Kong
Other Study IDs: CRE-2022.361
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Chronic Kidney Disease stage4; Chronc Kidney Disease Stage 5
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — Nirmatrelvir-ritonavir (Paxlovid)
  Other Names: Paxlovid

SUMMARY:
Nirmatrelvir-ritonavir is approved for coronavirus disease 2019 (COVID-19) but not initially recommended in patients with severe renal impairment. Increasing observational data have shown the feasibility of dose-adjusted nirmatrelvir-ritonavir administration in patients with estimated glomerular filtration rate lower than 30 ml/min/1.73 m^2. The study is planned to assess the safety, clinical and virologic outcomes of early oral nirmatrevir-ritonavir treatment of COVID-19 in patients with stage 4 and 5 chronic kidney disease.

DETAILED DESCRIPTION:
The objectives of the study are to evaluate the safety and clinical and virologic outcomes of dose-adjusted nirmatrelvir-ritonavir in patients with eGFR lower than 30 ml/min/1.73 m^2. Patients with eGFR greater than 30 ml/min/1.73 m2 and prescribed nirmatrelvir-ritonavir will be used for comparison.

In the single-centre study, patients with stage 4 and 5 chronic kidney disease prescribed early treatment dose-adjusted nirmatrelvir-ritonavir will be assessed for the primary endponts of adverse events during or after treatment with nirmatrelvir-ritonavir (starting on or before day 30), serious adverse events and adverse events leading to discontinuation of nirmatrelvir-ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above.
* COVID-19 infection and symptom onset no more than 5 days, with or without prior vaccination.
* WHO CPS 1-4
* Indicated for nirmatrelvir-ritonavir treatment

Exclusion Criteria:

* Patients cannot swallow capsules or adhere to protocol.
* Severe COVID-19 disease, including patients who require oxygen supplement therapy
* Significant hypersensitivity to nirmatrelvir, ritonavir, or any component of the formulation
* Patients require co-administration of drugs that are highly dependent on CYP3A4 for clearance and cannot be omitted during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single centre study of 100 adult patients treated with nirmatrelvir-ritonavir for early COVID-19 disease in the omicron era.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
adverse event | 30 days
  Adverse events during or after treatment with nirmatrelvir-ritonavir (starting on or before day 30), serious adverse events and adverse events leading to discontinuation of nirmatrelvir-ritonavir

SECONDARY OUTCOMES:
RAT | 30 days
  Time to negative rapid antigen test result
Rebound | 30 days
  Rebound of positive rapid antigen test or polymerase chain reaction PCR up to day 30
WHO Clinical Progression Scale CPS | 30 days
  Time to progression to CPS 5 up to day 30
Symptoms | 30 days
  Time to resolution of symptoms
Symptomatic rebound | 30 days
  Symptomatic rebound (symptomatic again after resolution of symptom with positive RAT or PCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan GCK, Lui GCY, Wong CNS, Yip SST, Li TCM, Cheung CSK, Sze RKH, Szeto CC, Chow KM. Safety Profile and Clinical and Virological Outcomes of Nirmatrelvir-Ritonavir Treatment in Patients With Advanced Chronic Kidney Disease and Coronavirus Disease 2019. Clin Infect Dis. 2023 Nov 17;77(10):1406-1412. doi: 10.1093/cid/ciad371. PMID 37531093